CLINICAL TRIAL: NCT03688412
Title: RELEASE: Transvenous Lead Removal Using the Cook Evolution® Lead Extraction System Post-Market Clinical Study.
Brief Title: Transvenous Lead Removal Post-Market Clinical Study
Status: Completed | Type: Observational
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Other Study IDs: 16-04
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Cardiac Electrophysiology
Keywords: Cardiac pacing, artificial; Cardiac Resynchronizaton Therapy Devices; Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cook lead extraction devices: The Cook lead extraction devices are indicated for use in patients requiring percutaneous removal of CIED leads, indwelling catheters and foreign objects.
  Interventions: Device: Cook lead extraction devices

INTERVENTIONS:
Device: Cook lead extraction devices — The Cook lead extraction devices are mechanical devices that encompass a full variety of devices required for percutaneous removal of CIED leads, indwelling catheters and foreign objects.

SUMMARY:
This prospective, multicenter, post-market clinical study was designed to evaluate the outcomes of lead extraction of cardiovascular implantable electronic devices (CIED) using Cook catheter and lead extraction devices for any indication it is used in the commercial setting within the United States and Europe. The purpose of this clinical study is to collect data on the performance of the Cook lead extraction devices for the purpose of supporting publications and presentations

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age or older
2. Lead indwell time greater than 1 year

Exclusion Criteria:

1. Patient is unable or unwilling to provide informed consent (per the IRB/EC requirements) to participate in the clinical study
2. Patient presents with an extracardiac lead

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients requiring percutaneous removal of Cardiovascular Implantable Electronic Device (CIED) leads
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-05-11 (Actual)

PRIMARY OUTCOMES:
Rate of complete procedural success | Immediately following lead extraction
  Complete procedural success is the removal of the targeted lead and all lead material from the vascular space, with the absence of permanently disabling complications or procedure-related death.
Rate of clinical procedural success | Immediately following lead extraction
  Clinical procedural success is the removal of all targeted leads and all lead material from the vascular space, or retention of a small portion of the lead (fragment that is 4 cm or smaller) that does not negatively impact the outcome goals of the procedure.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (6):
  - UCSF Medical Center, San Francisco, California
  - Carle Foundation, Urbana, Illinois
  - NC Heart and Vascular Reseach, Raleigh, North Carolina
  - Wellspan York Hospital, York, Pennsylvania
  - Memorial Hermann, Houston, Texas
  - University of VA Medical Center, Charlottesville, Virginia
- German Heart Center Berlin, Berlin, Germany
- Isala, Zwolle, Netherlands
- St. George's University Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Cook Research Incorporated (CRI) is fully committed to supporting the principles of responsible data sharing, including providing qualified scientific researchers access to deidentified, patient-level data from CRI clinical studies to conduct legitimate scientific research. Data underlying the results reported in this clinical study will be made available for request after publication of the results from this study and ending 5 years after initial publication. Interested researchers may review the "Cook Research Incorporated Policy on Access to Clinical Study Data" at https://www.cookresearchinc.com/extranet/data-access.html and submit a complete research proposal to request data access. Additional study documents (such as the study protocol) will be shared as needed if the data access request is granted. A data sharing agreement will be executed for access to deidentified patient-level data.